CLINICAL TRIAL: NCT01558765
Title: CopenHeartVR - A Randomized Clinical Trial Investigating the Effect of Integrated Rehabilitation Versus Usual Care Without Physical Exercise After Heart Valve Surgery.
Brief Title: CopenHeartVR - Integrated Rehabilitation of Patients After Heart Valve Surgery
Acronym: CopenHeartVR
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Selina Kikkenborg Berg, Principal Investigator, RN, MSN, PhD, FESC., Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RHCopenHeartVR
Record Dates: First submitted 2012-03-16; First posted 2012-03-20 (Estimated); Last update posted 2015-11-13 (Estimated); Status verified 2015-11

CONDITIONS: Heart Valve Disease
Keywords: Rehabilitation; Integrated rehabilitation programme; Exercise training; Psycho-educational care
MeSH Terms: conditions — Heart Valve Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention group (Experimental): Patients receive integrated rehabilitation
  Interventions: Other: Integrated rehabilitation
- Control group (No Intervention): Patients receive usual follow-up care without physical exercise

INTERVENTIONS:
Other: Integrated rehabilitation — Integrated rehabilitation consisting of exercise training (3 times per week (1 hour) for 12 weeks) and psycho-educational care (5 consultations over 6 months by special trained nurses).
  Arms: Intervention group

SUMMARY:
The aim of the study is to investigate the effect of an integrated rehabilitation programme, consisting of physical exercise training and psycho-educational consultations, for patients after heart valve surgery.

The hypothesis is that integrated rehabilitation can improve physical capacity measured by V02 peak, self-rated mental health and life quality by validated questionnaires such as SF-36, and other objective parameters such as cardiac-specific biomarkers and echocardiographic measurements.

DETAILED DESCRIPTION:
Worldwide, the incidence of heart valve disease is increasing. Improved surgical techniques, rising age and possibility for re-operation leads to a rising number of patients having heart valve surgery. The gap between hospital discharge and returning to normal life is obvious. Integrated rehabilitation could probably reduce hospital readmissions, increase physical capacity and increase self-rated mental health and quality of life. Therefore the aim of this study is to explore if patients after heart valve surgery will benefit from an integrated rehabilitation programme consisting of physical exercise and psycho-educational intervention.

A randomized clinical trial is conducted to investigate the effect and meaning of an integrated rehabilitation programme on the physical and psychosocial functioning of patients after heart valve surgery. The trial is a parallel arm design.

A mixed methods embedded experimental design is chosen to include both quantitative and qualitative data to evaluate the intervention. The intervention consists of five psycho-educational consultations provided by specialized nurses and a twelve week individualized exercise training programme provided by physiotherapists. A qualitative post-intervention study will explore rehabilitation participation experiences.

Along with the above stated hypothesis, it will be observed whether integrated rehabilitation can reduce anxiety, depression, health care utilisation, mortality and work cessation.

210 patients will be included.

Validated questionnaires (e.g. SF-36), cardiopulmonary exercise testing, 6 minute walking test, echocardiography, cardiac-specific biomarkers and qualitative interviews will be used to evaluate the effect and meaning of the programme.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to hospital for elective heart valve surgery at Rigshospitalet, Denmark
* 18 years or older
* Speak and understand Danish
* Providing written informed consent

Exclusion Criteria:

* Known ischemic heart disease prior to heart valve surgery
* Is included in an other clinical trial investigating the effects of physical training and psycho-educational intervention
* Unable to understand and cooperate to study instructions
* Pregnant and/or breast feeding
* Performing exercise training at high level and several times a week
* No written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 147 (Actual)
Dates: Start 2012-03; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Change in physical capacity | 1,4,12 months
  Measured by Vo2peak by ergospirometry testing

SECONDARY OUTCOMES:
Change in self-rated mental health and quality of life | 0, 1, 4, 6, 12 and 24 months
  Measured by total score and the mental health component scale (MSC) in the SF-36 questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Kirstine Laerum Sibilitz, MD, Principal Investigator — Rigshospitalet, Denmark; Ann-Dorthe Zwisler, MD, Ph.d., Principal Investigator — Rigshospitalet / Copenhagen University Hospital, National Institute of Public Health, University of Southern Denmark; Selina Kikkenborg Berg, Ph.d., Principal Investigator — Rigshospitalet, Denmark; Christian Hassager, MD, DMSc, Principal Investigator — Rigshospitalet, Denmark; Lars Køber, MD, DMSc, Principal Investigator — Rigshospitalet, Denmark; Daniel Steinbrüchel, MD, DMSc, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet / Copenhagen University Hospital, Copenhagen, Copenhagen, Denmark

REFERENCES:
- [Derived] Sibilitz KL, Berg SK, Rasmussen TB, Risom SS, Thygesen LC, Tang L, Hansen TB, Johansen PP, Gluud C, Lindschou J, Schmid JP, Hassager C, Kober L, Taylor RS, Zwisler AD. Cardiac rehabilitation increases physical capacity but not mental health after heart valve surgery: a randomised clinical trial. Heart. 2016 Dec 15;102(24):1995-2003. doi: 10.1136/heartjnl-2016-309414. Epub 2016 Aug 4. PMID 27492941
- [Derived] Sibilitz KL, Berg SK, Hansen TB, Risom SS, Rasmussen TB, Hassager C, Kober L, Gluud C, Thygesen LC, Lindschou J, Schmid JP, Taylor RS, Zwisler AD. Update to the study protocol, including statistical analysis plan for a randomized clinical trial comparing comprehensive cardiac rehabilitation after heart valve surgery with control: the CopenHeartVR trial. Trials. 2015 Feb 5;16:38. doi: 10.1186/s13063-015-0562-z. PMID 25887433
- [Derived] Sibilitz KL, Berg SK, Hansen TB, Risom SS, Rasmussen TB, Hassager C, Kober L, Steinbruchel D, Gluud C, Winkel P, Thygesen LC, Hansen JL, Schmid JP, Conraads V, Brocki BC, Zwisler AD. Effect of comprehensive cardiac rehabilitation after heart valve surgery (CopenHeartVR): study protocol for a randomised clinical trial. Trials. 2013 Apr 22;14:104. doi: 10.1186/1745-6215-14-104. PMID 23782510